CLINICAL TRIAL: NCT06839768
Title: The MILES Trial: Prospective Randomized Trial of Safety and Efficacy of Minimally-invasive Versus Standard Laser Enucleation of the Prostate
Brief Title: Safety and Efficacy of MILEP Versus Standard EEP
Acronym: MILES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sechenov University (Other)
Collaborators: Hospital Pompeia (Other)
Responsible Party: Principal Investigator, Vladislav Petov, Assosiate Professor, urologist, Sechenov University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MILEP2024_0.1
Record Dates: First submitted 2025-01-13; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Benign Prostate Hypertrophy(BPH); LUTS(Lower Urinary Tract Symptoms)
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MiLEP (22 Ch) (Experimental)
  Interventions: Procedure: MiLEP
- EEP (26 Ch) (Active Comparator)
  Interventions: Procedure: Standard endoscopic enucleation of the prostate (EEP)

INTERVENTIONS:
Procedure: Standard endoscopic enucleation of the prostate (EEP) — Stabdard EEP will be nerformed using 26 Ch resectoscope. Enucleation will be performed using an en bloc no-touch technique with early apical release.
  Arms: EEP (26 Ch)
Procedure: MiLEP — Minimally-invasive laser EEP will be nerformed using 22 Ch resectoscope. Enucleation will be performed using an en bloc no-touch technique with early apical release.
  Arms: MiLEP (22 Ch)

SUMMARY:
Endoscopic enucleation of the prostate (EEP) is a standard treatment for benign prostatic hyperplasia (BPH), with modifications such as MiLEP that utilizes smaller instruments. The reduced resectoscope diameter in MiLEP may help decrease rates of stress urinary incontinence (SUI) and urethral strictures.

Objective: to compare the efficacy and safety of MiLEP and standard EEP with a thulium fiber laser (TFL).

ELIGIBILITY:
Inclusion Criteria:

LUTS presence, proven by:

1. IPSS questionnaire (Score >20);
2. OR uroflowmetry result (Qmax <10 ml/s);

Exclusion Criteria:

* Prostate volume > 120 cc
* Prostate cancer on pathology;
* Urethral strictures;
* Bladder calculi;
* Prior prostate surgery;
* Neurogenic bladder dysfunction.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
The rate of SUI | 1 month

SECONDARY OUTCOMES:
Rate of urethral strictures | 6-12 months
Rate of intra- and perioperative adverse events | the day of operation, at 1, 6,12 months post-operative
  Assessed using Clavien-Dindo classification system
Operative time | participants will be followed for the duration of the intervention, an expected average of 1 hour
Blood loss (blood levels of haemoglobin and haematocrit) | 1 day before and 1 day after surgery
Catheterization time | participants will be followed for the duration of hospital stay, an expected average of 1,5 days
Hospital stay | participants will be followed for the duration of hospital stay, an expected average of 1,5 days
International Prostate Symptom Score (IPSS) | 1 month
  Mild LUTS (symptom score less than of equal to 7) Moderate LUTS (symptom score range 8-19) Severe LUTS (symptom score range 20-35)
Qmax | 1 month
PVR | 1 month
International Index of Erectile Function (IIEF-5) | 1 month
  severe ED (5-7), moderate ED (8-11), mild to moderate ED (12-16), mild ED (17-21), and no ED (22-25)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Urology and Reproductive Health, Sechenov University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No